CLINICAL TRIAL: NCT04758013
Title: Comparison of Changes of ONSD Between Groups of Laparoscopic Surgery With and Without Epidural Saline Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Seob Kim, Assistant Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KeimyungUniversity
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Optic Nerve Sheath Diameter; Pneumoperitoneum; Epidural
Keywords: ONSD; pneumoperitoneum; epidural
MeSH Terms: conditions — Pneumoperitoneum | interventions — Injections, Epidural

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laparoscopic gastric surgery with Epidural injection (Experimental): Patients with laparoscopic gastric surgery who received epidural injection through an thoracic epidural catheter.
  Interventions: Procedure: Epidural injection through thoracic epidural catheter
- Laparoscopic gastric surgery without Epidural injection (Experimental): Patients with laparoscopic gastric surgery who don't received epidural injection through an thoracic epidural catheter.
  Interventions: Procedure: Without epidural injection
- Open gastric surgery (No Intervention): Patients with open gastric surgery.

INTERVENTIONS:
Procedure: Epidural injection through thoracic epidural catheter — The investigators inject drugs through a catheter inserted into the thoracic epidural space to control pain after surgery in patients undergoing gastric surgery by laparoscopy.
  Arms: Laparoscopic gastric surgery with Epidural injection
Procedure: Without epidural injection — The investigators don't epidural injection to find out the effect of only inter-abdominal pressure on intracranial pressure.
  Arms: Laparoscopic gastric surgery without Epidural injection

SUMMARY:
This study targets patients undergoing laparoscopic gastric cancer surgery.

The investigators would like to compare two factors that influence intracranial pressure through optic nerve sheath diameter measurement.

First factor is intraperitoneal pressure.

Second factor is epidural pressure.

The investigators divided the patients into three groups.

Group A is patients with laparoscopic gastric surgery who received epidural injection through an thoracic epidural catheter.

Group B is patients with laparoscopic gastric surgery who don't received epidural injection through an thoracic epidural catheter.

Group C is patients with open gastric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Gastric surgery due to cancer

Exclusion Criteria:

* Coagulopathy
* Infection
* Previous history of thoracic spine surgery
* Ophthalmic diseases
* History of increased Intracranial Pressure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-16 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
T0 : Optic nerve sheath diameter | 10 minutes after anesthesia induction
  The investigator measures Optic nerve sheath diameter by ultrasonography.
T1 : Optic nerve sheath diameter | 10min after entering the laparoscope
  The investigator measures Optic nerve sheath diameter.
T2 : Optic nerve sheath diameter | 1hour after entering the laparoscope
  The investigator measures Optic nerve sheath diameter.
T3 : Optic nerve sheath diameter | 10min after the laparoscopy comes out
  The investigator measures Optic nerve sheath diameter.

CONTACTS AND LOCATIONS:
Overall Officials: JiSeob Kim, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- KeimyungUniversity, Daegu, South Korea

REFERENCES:
- [Derived] Kim JS, Hong JH, Park JH. Comparison of Changes in the Optic Nerve Sheath Diameter Following Thoracic Epidural Normal Saline Injection in Laparoscopic Surgery. Pain Physician. 2022 Jul;25(4):E563-E569. PMID 35793180